CLINICAL TRIAL: NCT01484158
Title: Gait Speed for Predicting Cardiovascular Events After Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Principal Investigator, Yasushi Matsuzawa, Primary Investigator, Yokohama City University Medical Center
Other Study IDs: Gait Speed Outcome Study
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We retain only blood sample only in this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myocardial Infarction: Patients with myocardial infarction

SUMMARY:
There are growing evidences that gait speed is inversely associated with all causes mortality especially cardiovascular mortality among the elderly. The purpose of this study is to evaluate the predictive value of gait speed for cardiovascular events in patients after ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
The investigators will enroll patients capable of walking with STEMI. All patients will receive successful reperfusion therapy within 12-hour from onset. Gait speed during cardiac rehabilitation is measured. Cardiovascular events were defined as a composite of cardiovascular death, non-fatal myocardial infarction and non-fatal stroke, for an average follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ST-segment elevation acute myocardial infarction
* Must be treated within 12 hours after symptom onset
* Must be able to walk
* Must receive successful primary percutaneous coronary intervention

Exclusion Criteria:

* History of prior myocardial infarction
* Cerebrovascular disease with residual hemiplegia
* Severe peripheral arterial disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2001-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Events | 5 years
  cardiovascular death, non-fatal myocardial infarction and non-fatal stroke

REFERENCES:
- [Derived] Matsuzawa Y, Konishi M, Akiyama E, Suzuki H, Nakayama N, Kiyokuni M, Sumita S, Ebina T, Kosuge M, Hibi K, Tsukahara K, Iwahashi N, Endo M, Maejima N, Saka K, Hashiba K, Okada K, Taguri M, Morita S, Sugiyama S, Ogawa H, Sashika H, Umemura S, Kimura K. Association between gait speed as a measure of frailty and risk of cardiovascular events after myocardial infarction. J Am Coll Cardiol. 2013 May 14;61(19):1964-72. doi: 10.1016/j.jacc.2013.02.020. Epub 2013 Mar 14. PMID 23500222